CLINICAL TRIAL: NCT04815694
Title: THeragnostic Utilities for Neoplastic DisEases of the Rectum by MRI Guided Radiotherapy
Acronym: THUNDER2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Principal Investigator, Giuditta Chiloiro, Principal Investigator, Medical Doctor PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3460
Record Dates: First submitted 2021-03-12; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Neoadjuvant Chemoradiotherapy; Locally Advanced Rectal Cancer; Pathological Complete Response
Keywords: MRI guided radiotherapy; Early Regression Index- ERI

STUDY DESIGN:
Intervention Model Description: The initial radiotherapy treatment will consist in delivering 55 Gy in 25 fractions on GTV plus the corresponding mesorectum of 45Gy in 25 fractions on the whole pelvis. Chemotherapy with 5-fluorouracil (5-FU) or oral capecitabine will be administered continuously. A 0.35 Tesla Magnetic resonance image will be acquired at simulation and every day during MRgRT. At fraction 10, ERI will be calculated. If ERI will be inferior than 13.1 the patient will continue the original treatment. If ERI will be higher than 13.1 the treatment plan will be reoptimized considering the residual tumor at fraction 10 as new therapy volume, where the dose will be intensified to reach 60.1 Gy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LARC patients treated by MRgRT with Early Regression Index (ERI) at 10th fraction >13.1 (Experimental): All patients will be treated on MRgRT, at the second week , patients with an ERI > 13.1 will underwent RT dose intensification on GTV + 3 mm to 60.1 Gy with a Simultaneous Integrated Boost (SIB).
  Interventions: Radiation: RT Dose escalation in LARC patients with an Early Regression Index > 13.1 at second week on nCRT
- LARC patients treated by MRgRT with Early Regression Index (ERI) at 10th fraction < 13.1 (No Intervention): All patients will be treated on MRgRT, at the second week , patients with an ERI < 13.1 will underwent standard RT dose of 55Gy on tumor and corresponding mesorectum

INTERVENTIONS:
Radiation: RT Dose escalation in LARC patients with an Early Regression Index > 13.1 at second week on nCRT — The initial radiotherapy treatment will consist in delivering 55 Gy in 25 fractions on GTV plus the corresponding mesorectum of 45Gy in 25 fractions on the whole pelvis. Chemotherapy with 5-fluorouracil (5-FU) or oral capecitabine will be administered continuously. A 0.35 Tesla Magnetic resonance image will be acquired at simulation and every day during MRgRT. At fraction 10, ERI will be calculated. If ERI will be inferior than 13.1 the patient will continue the original treatment. If ERI will be higher than 13.1 the treatment plan will be reoptimized considering the residual tumor at fraction 10 as new therapy volume, where the dose will be intensified to reach 60.1 Gy.
  Arms: LARC patients treated by MRgRT with Early Regression Index (ERI) at 10th fraction >13.1

SUMMARY:
Neoadjuvant chemoradiation therapy (nCRT) is the standard treatment modality in locally advanced rectal cancer (LARC) and patients achieving complete response to treatment (CR) usually have a better prognosis in terms of local control (LC), metastases-free survival (MFS) and overall survival (OS).

Recently, an early tumour regression index (ERITCP) was introduced, to predict pathological CR (pCR) after nCRT in LARC patients. In particular, the authors found that the patients with ERITCP <13.1 show a strong response during therapy and have a lower probability to experience distant relapses.

Aim of this clinical trial is to investigate the impact of dose escalation in rectal cancer, identifying the poor responder cases using the ERI index during the course of radiotherapy and increasing the prescribed dose in these patients.

Adopting this boosting protocol, an increase of 10% of CR (clinical and pathological) rate is expected.

For patients enrolled in the trial, chemoradiotherapy (CRT) will be administered using the MRI guided Radiotherapy (MRgRT) machine available in our institution.

If ERI will be inferior than 13.1 the patient will continue the original treatment. Patients with complete clinical response will go through wait and see approach.

If ERI will be higher than 13.1 the treatment plan will be reoptimized considering the residual tumor at fraction 10 as new therapy volume, where the dose will be intensified to reach 60.1 Gy.

The number of cases to be enrolled will be 63. The primary endpoints will be complete response considered as: ypT0N0 in case of Total Mesorectal Excision (TME), ypT0ycN0 in case of LE, ycT0N0 in case of WW; prospective validation of delta radiomics MR-guide Radiotherapy model.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiation therapy (nCRT) is the standard treatment modality in locally advanced rectal cancer (LARC) and patients achieving complete response to treatment (CR) usually have a better prognosis in terms of local control (LC), metastases-free survival (MFS) and overall survival (OS).

Since response to radiotherapy is dose dependent in rectal cancer, dose escalation may lead to higher complete response rates. The possibility to predict patients who will achieve CR before surgery or during nCRT is of crucial importance. Recently, an early tumour regression index (ERITCP) was introduced, to predict pathological CR (pCR) after nCRT in LARC patients. In particular, the authors found that the patients with ERITCP <13.1 show a strong response during therapy and have a lower probability to experience distant relapses.

Aim of this clinical trial is to investigate the impact of dose escalation in rectal cancer, identifying the poor responder cases using the ERI index during the course of radiotherapy and increasing the prescribed dose in these patients.

Adopting this boosting protocol, an increase of 10% of CR (clinical and pathological) rate is expected.

For patients enrolled in the trial, chemoradiotherapy (CRT) will be administered using the MRI guided Radiotherapy (MRgRT) machine available in our institution.

The initial radiotherapy treatment will consist in delivering 55 Gy in 25 fractions on Gross Tumor Volume (GTV) plus the corresponding mesorectum of 45Gy in 25 fractions on the whole pelvis. Chemotherapy with 5-fluorouracil(5-FU) or oral capecitabine will be administered continuously.

A 0.35 Tesla Magnetic Resonance image will be acquired at simulation and every day during MRgRT. At fraction 10, ERI will be calculated.

If ERI will be inferior than 13.1 the patient will continue the original treatment. Patients with complete clinical response will go through wait and see approach.

If ERI will be higher than 13.1 the treatment plan will be reoptimized considering the residual tumor at fraction 10 as new therapy volume, where the dose will be intensified to reach 60.1 Gy.

After the end of CRT, the clinical response will be evaluated 8-10 weeks using high tesla MR and CT images or FDGPET-CT image 8-10 weeks after the end of nCRT. Surgery will be performed 12-16 weeks after the end of the CRT in case of partial or stable or progression disease, while in case of major or complete clinical response at restaging imaging, a Watch and Wait (W&W) or local excision (LE) approach should be followed. Late toxicity and quality of life (QoL) will be scored at first follow-up (FUP) and at 1 and 2 years of FUP according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0 scale, functional scales and QoL questionnaires (LARS and SEXUAL questionnaires, at the start of treatment, after surgery and at 1 and 2 years of FUP), respectively.

The number of cases to be enrolled will be 63: all the patients will be treated at Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome. All the cases will be discussed in weekly multidisciplinary tumor board to share the best therapeutic options, both at the diagnosis and at presurgical restaging.

. The primary endpoints will be complete response considered as: ypT0N0 in case of Total Mesorectal Excision (TME), ypT0ycN0 in case of LE, ycT0N0 in case of WW; prospective validation of delta radiomics MR-guide Radiotherapy model.

The secondary endpoints will be:3 years LC, MFS, Disease Free Survival (DFS), OS; R0 resection rate; Tumor Regression Grade (TRG) 1, TRG 2, Neoadjuvant Rectal (NAR) score; Sphincter preservation rate; Organ preservation rate; Rectal and sexual functions.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven adenocarcinoma of the rectum cT2-3, N0-2 or cT4 for anal sphincter involvement N0-2a, M0
* No prior radiotherapy in pelvic region;
* Tumour located between 0 and 15 cm above the anal verge;
* Not mesorectal fascia involvement for tumor
* No extramesorectal nodes involvement
* No extramural venous invasion (EMVI)
* No rectal mucinous adenocarcinoma histology
* No contra-indications for MRI
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Age over 18 years
* Adequate hematological function: granulocyte count > 1500/microl; Hemoglobin level > 10 g/dl; Platelet count > 100000/microl; Alanine Aminotransferase/ aspartate aminotransferase (ALT/AST): 7-45 UI/L;
* No other malignancies in the previous history (except skin and initial cervical cancer);
* Absence of important comorbidities: severe cardiac or coagulative disease, moderate or severe; restrictive/obstructive lung deficit, severe cognitive impairment, moderate and severe renal and hepatic impairment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Absence of pregnancy or lactating female patients;
* Written informed consent

Exclusion Criteria: not defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete response | 6 months
  ypT0N0 in case of TME, ypT0ycN0 in case of LE, ycT0N0 in case of WW
Prospective validation of delta radiomics MR-guide Radiotherapy model | 6 months
  correlation between response prediction and clinical or pathological response

SECONDARY OUTCOMES:
3 years Local control | 3 years follow up
  survival outcomes
3 years Metastasis Free Survival | 3 years follow up
  survival outcomes
3 years Disease Free Survival | 3 years follow up
  survival outcomes
3 years Overall Survival | 3 years follow up
  survival outcomes
R0 resection rate | 6 months
  percentage of surgical intervention with negative margins
Tumor Regression Grade 2 | 6 months
  surgical outcomes
Neoadjuvant rectal (NAR) score | 6 months
  surgical outcomes
Tumor Regression Grade 1 | 6 months
  surgical outcomes
Sphincter preservation rate | 6 months
  percentage of surgical intervention without the positioning of permanent stomia
Organ preservation rate | 3 years follow up
  percentage of patients underwent conservative approaches (WW or EL)
Rectal function | 3 years follow up
  impact of therapy on rectal functions by MSKCC questionnaire (from always to never with 5 items)
Sexual function | 3 years follow up
  impact of therapy on sexual function by IIEF and FSFI questionnaires (from 1 worst to 5 better)

CONTACTS AND LOCATIONS:
Overall Officials: Giuditta Chiloiro, MD PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiloiro G, Cusumano D, Boldrini L, Romano A, Placidi L, Nardini M, Meldolesi E, Barbaro B, Coco C, Crucitti A, Persiani R, Petruzziello L, Ricci R, Salvatore L, Sofo L, Alfieri S, Manfredi R, Valentini V, Gambacorta MA. THUNDER 2: THeragnostic Utilities for Neoplastic DisEases of the Rectum by MRI guided radiotherapy. BMC Cancer. 2022 Jan 15;22(1):67. doi: 10.1186/s12885-021-09158-9. PMID 35033008

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04815694/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04815694/ICF_001.pdf